CLINICAL TRIAL: NCT05627700
Title: A Prospective, Open-label, Single-center Study of the Atia™ AVL200 Modular Intraocular Lens System for Treatment of Cataract and Presbyopia
Brief Title: AVL200 IOL for Treatment of Cataract and Presbyopia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atia Vision (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP100962
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- AVL200 IOL (Experimental): The AVL200 is a modular fluid-filled, shape-changing intraocular lens (IOL) designed to restore visual function across a range of focal points
  Interventions: Device: AVL200 IOL

INTERVENTIONS:
Device: AVL200 IOL — The AVL200 is an intraocular lens surgically implanted in the eye after cataract surgery.

SUMMARY:
This study is to evaluate the performance of the AVL200 IOL in terms of visual function improvement over a range of focal points. Participants meeting eligibility criteria will undergo cataract surgery with implantation of the AVL200 intraocular lens (IOL), then be followed through 1 year postoperatively. Postoperative assessments include safety and visual function.

ELIGIBILITY:
Inclusion Criteria:

* Visually significant cataract
* Best corrected distance visual acuity between 20/40 and 20/200
* Potential distance visual acuity of 20/32 or better
* Corneal astigmatism ≤ 1.5 diopters

Exclusion Criteria:

* Use of medication that could affect accommodation
* Previous corneal surgery or significant corneal abnormalities
* Ocular pathology or degenerative disorder having potential to impair visual acuity
* Pupil abnormality
* Intraoperative cataract surgery complications that could affect IOL implantation or positioning

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in monocular best corrected distance visual acuity | 3 months postoperative
  Best-corrected distance visual acuity as measured using an early-treatment diabetic retinopathy study (ETDRS) eye chart

SECONDARY OUTCOMES:
Change in monocular distance-corrected near visual acuity | 3 months postoperative
  Distance-corrected distance visual acuity as measured using an early-treatment diabetic retinopathy study (ETDRS) eye chart

CONTACTS AND LOCATIONS:
Overall Officials: Ashvin Agarwal, MD, Principal Investigator — Dr. Agarwals Eye Hospital
Locations (1):
- Dr Agarwal's Eye Hospital, Chennai, Tamal Nadu, India

IPD SHARING:
Plan to Share IPD: No